CLINICAL TRIAL: NCT06206928
Title: Investigation of Trace Element Metabolism and Tricarboxylic Acid Cycle Enzyme Activities in Patients Who Underwent Cesarean Section With Spinal Anesthesia
Brief Title: Evaluation of Mitochondrial Enzyme Activity in Cesarean Section Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Tercan, Associate professor, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: HRÜ/22.15.11
Record Dates: First submitted 2023-12-27; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Cesarean Section; Spinal Anesthesia; Thiol Groups
Keywords: cesarean section; spinal anesthesia; mitochondrial enzyme changes; thiol disulfide balance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about in effects of trace element metabolism, tricarboxylic acid cycle enzyme activities and thiol/disulfide balance in patients who underwent cesarean section under spinal anesthesia. The main question[s] it aims to answer are:

• What is the effect of trace element metabolism, tricarboxylic acid cycle enzyme activities and thiol/disulfide balance in patients undergoing cesarean section under regional anesthesia? A 10 ml blood sample will be taken from the participants to analyze the biochemical parameters mentioned before and after the operation. Pre- and post-operative values will be compared.

DETAILED DESCRIPTION:
Although the World Health Organization recommends the cesarean birth rate as 10-15%, the cesarean birth rate in Turkey is 57.3% according to 2020 data, ranking first in the world. This rate is around 30% for primary cesarean delivery. Although there are various methods of anesthesia for cesarean birth, spinal block is a regional anesthesia method frequently used in elective cesarean births because it is easy to apply, has a rapid onset of effect and provides a good sensory block. With this anesthesia method, local anesthetic solution is administered to the subarachnoid space to create sensory and motor block within the surgical area.

Although trace elements (Zinc (Zn), Iron (Fe), Copper (Cu)) constitute a small part of the human body, they play a very important role in maintaining normal metabolic function. Deficiency or excess of these elements causes dysfunction of the relevant enzymes (such as alcohol dehydrogenase, alkaline phosphatase, lactate dehydrogenase, carboxypeptidase, carbonic anhydrase, superoxide dismutase (SOD), DNA and RNA polymerase) and thus various clinical findings (postpartum hemorrhage, fetal growth restriction). FGR), fetal malformations, premature birth, preeclampsia).

In recent years, it has been revealed that thiol-disulfide homeostasis may be an important biomarker of oxidative stress. Thiol is a compound containing sulfhydryl group (-SH) that plays an important role in preventing oxidative stress in cells. Thiols are not only a redox buffer in the body but also an essential element of the antioxidant defense system. Abnormal thiol-disulfide balance levels are associated with oxidative stress. There is a balance between oxidative stress and antioxidant defense mechanisms. The changes in this balance depending on many factors are frequently investigated in patients undergoing surgery.

This study aimed to contribute to the literature by investigating the effects of trace element metabolism, tricarboxylic acid cycle enzyme activities and thiol/disulfide balance in patients who underwent cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo planned cesarean section between the ages of 18 and 40
2. ASA 1-2 Patients

Exclusion Criteria:

1. Patients who refuse to participate in the study
2. Patients over 40 years of age
3. ASA 3-4 Patients
4. Patients who underwent emergency cesarean section
5. Those with known liver and kidney diseases, patients diagnosed with Diabetes Mellitus
6. Pregnant women diagnosed with an abnormal baby
7. Patients diagnosed with preeclampsia
8. Patients with body mass index ≥ 30
9. Patients who do not accept spinal anesthesia or have contraindications to the application -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since this study was planned in patients who underwent cesarean section under spinal anesthesia
Study Population: Patients who will undergo planned cesarean section between the ages of 18 and 40
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical parameter measurements that we mentioned in the description | 1 day
  Serum zinc concentrations were measured with commercially available Rel Assay zinc measurement kit (Gaziantep, Turkey) using a fully automatic photometric method (Abbott ARCHITECT c8000 clinical chemistry analyzer).
  Serum copper concentrations were measured with commercially available Rel Assay copper measurement kit (Gaziantep, Turkey), using a fully automatic photometric method (Abbott ARCHITECT c8000 clinical chemistry analyzer).
  Serum levels of total and native thiol were measured with a novel method developed by Erel and Neselioglu. In this method, serum dynamic disulfide bonds (-S-S-) is reduced to native thiol groups (-SH HS-) by sodium borohydride (NaBH4) and native thiol levels were measured.

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET TERCAN, Assoc Prof, Principal Investigator — University of Health science
Locations (1):
- Şanlıurfa Training and Research Hospital, Sanliurfa, Turkey (Türkiye)